CLINICAL TRIAL: NCT00365040
Title: Customized PRK With Mitomycin Versus Customized Lasik for Myopic Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AWMC
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2006-08-17 (Estimated); Status verified 2006-07

CONDITIONS: Refractive Errors
Keywords: myopia; excimer laser
MeSH Terms: conditions — Refractive Errors; Myopia | interventions — Photorefractive Keratectomy

INTERVENTIONS:
Procedure: Prk with mitomycin vs Lasik

SUMMARY:
The present study was designed to compare the use of mitomycin in PRK for the treatment of refractive errors and to compare these results to customized Lasik

ELIGIBILITY:
Inclusion Criteria:

* Myopia or compound myopic astigmatism, stable refractive error, no associated eye disease

Exclusion Criteria:

* Diabetes, autoimmune diseases, topographic abnormalities

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-12; Study Completion 2006-10

PRIMARY OUTCOMES:
visual acuity
refractive errors
topography patterns
aberrometry data

SECONDARY OUTCOMES:
subjective evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Campos, MD, Study Chair — Federal University of São Paulo